CLINICAL TRIAL: NCT02647502
Title: A Pilot Study of Intermittent Calorie Restriction in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Ellen M. Mowry, Associate Professor of Neurology and Epidemiology, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00065806
Record Dates: First submitted 2015-12-28; First posted 2016-01-06 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Continuous calorie restriction (Active Comparator): Participants will be provided with a diet that includes approximately 78% of calories each day that would be needed to maintain current BMI.
  Interventions: Other: Diet
- Intermittent calorie restriction (Experimental): Participants will be provided a diet that with a daily calorie intake required to maintain current BMI, except only 25% of this calorie intake will be provided for 2 days a week.
  Interventions: Other: Diet
- Control calorie intake (Placebo Comparator): Participants will be assigned to consume enough calories each day required to maintain current BMI
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Diet, standardized to the 50th percentile for macronutrients, will be provided at varied calorie levels as described.

SUMMARY:
Experimental studies of the experimental autoimmune encephalomyelitis (EAE), a mouse model of multiple sclerosis, indicate that the number of calories fed to mice prevent EAE and are also associated with less severe disease in mice who do develop the disease. Currently, whether these results translate favorably in humans is unknown. This is a pilot trial of testing two caloric restriction (CR) diets versus a control diet in multiple sclerosis (MS) patients: one continuous caloric restriction (CR) diet where a small number of calories will be restricted every day or another intermittent CR diet where a caloric intake will be restricted more severely 2 days per week. Participants are randomized to one of the diets, and for the first 8 weeks, will receive standardized, prepared meals tailored to the specific diet. At the conclusion of the controlled feeding study, all participants will transition to an unblinded phase for an additional 40 weeks where they are provided with instructions to follow an intermittent CR diet.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-50
* Capable of storing food safely, willing to follow diet/eat provided food, and able to receive shipments at home or work
* Meets 2010 criteria for McDonald MS;
* Relapse or new lesion in previous 2 years
* Expanded disability status score (EDSS) < 6
* Disease duration ≤15 years
* Untreated or on stable on first-line MS therapy [injectable] for at least 6 months, with no anticipated changes in the next 10 weeks
* Unchanged vitamin D dose or thyroid replacement dose (for those on it) with no anticipated changes or in supplement use for the next 10 weeks.
* Non-regular smoker (average no more than 1 cigarette/day) for at least 2 months
* Stable weight, by self report, for past 3 months (± 8 lbs)
* Body mass index (BMI) > 23 kg/m2

Exclusion Criteria:

* Pregnant or nursing, or unwilling to prevent pregnancy (if of childbearing to potential)

  * History of gastrointestinal disease causing malabsorption
  * History of diabetes requiring medication
  * History of stage IV/V chronic kidney disease or vascular disease
  * History of major surgery in past 3 months
  * Current use of warfarin
  * History of eating disorder
  * Currently on a special diet for MS/other diet (provided diet will be pork free)
  * Chemotherapy within the past year

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-12; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Adverse events | 8 weeks
  Adverse events will be categorized by organ system and by the blinded neurologist's assessment of the relation to the diet.

SECONDARY OUTCOMES:
Adherence to Calories Assigned | 8 weeks
  Adherence will be assessed by comparing the total caloric intake provided to the patients through the assigned diet to the total energy intake determined by the research dieticians.
Adherence to Calories Assigned | 48 weeks
  Adherence during the "advice-only" phase will be compared to adherence in each diet group during the first 8 weeks using paired t-tests, where the grouping is done naturally by subject.
Adverse Events | 48 weeks
  Adverse events will be categorized by organ system and by the blinded neurologist's assessment of the relation to the diet.
Quality of Life Questionnaire | 48 weeks
  "Functional Assessment in MS" results will be assessed during the study
NIH Patient-Reported-Outcomes Measurement Information System (PROMIS )Fatigue Questionnaire | 48 weeks
  PROMIS Fatigue results will be assessed during the study
Change in metabolite ratios | 8 weeks
  The impact of each calorie restriction diet versus control diet on the metabolomics profile will be assessed.
Immune cell subsets/cytokines | 8 weeks
  The impact of each calorie restriction diet versus control diet on ratios of immune cell subsets (e.g. T-helper (TH)17, TH1, TH2, T regulatory) and related cytokines will be assessed.
Change in concentration of measures of metabolism | 8 weeks
  The impact of each calorie restriction diet versus control diet on fasting glucose, insulin, leptin, ghrelin, C-reactive protein, lipids, and long-chain ceramides will be assessed.
Change in serum lipid concentration | 8 weeks
  The impact of each calorie restriction diet versus control diet on fasting lipids and long-chain ceramides will be assessed.
Change in serum brain-derived neurotrophic factor concentration (BDNF) | 8 weeks
  The impact of each calorie restriction diet versus control diet on fasting BDNF will be assessed.
Change in levels of oxidative stress biomarkers | 8 weeks
  The impact of each calorie restriction diet versus control diet on protein carbonyls, 8-isoprostane, nitrotyrosine, and 4-hydroxynonenal adducts will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Mowry, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States